CLINICAL TRIAL: NCT01136005
Title: Phase III Randomized Double-Blind Trial of Bepanthen® Cream Versus Cetomacrogol Cream in the Prevention of Papulopustular Eruption in Patients Receiving Epidermal Growth Factor Receptor Inhibitors (EGFRI): BeCet
Brief Title: Bepanthen Versus Cetomacrogol in Epidermal Growth Factor Receptor Inhibitors (EGFRI)
Acronym: BeCet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impaqtt Foundation (Other)
Collaborators: CB Boers ORG (Other); Memorial Sloan Kettering Cancer Center (Other); Leiden University Medical Center (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Impaqtt-001; M010-025 (Other: Medical research ethics committee: METC Noord Holland)
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer; Skin Rash
Keywords: receptor, epidermal growth factor; skin reactions; quality of life; adherence
MeSH Terms: conditions — Neoplasms; Exanthema | interventions — dexpanthenol; Provitamins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexpanthenol 5% cream (Experimental): dexpanthenol 5% cream
  Interventions: Other: dexpanthenol 5% cream
- cetomacrogol cream (Active Comparator): a vehicle
  Interventions: Other: Cetomacrogol cream

INTERVENTIONS:
Other: dexpanthenol 5% cream — Apply at least two times a day on face, chest and upper arms during the 6 week treatment period
  Other Names: Bepanthen; Provitamin
  Arms: dexpanthenol 5% cream
Other: Cetomacrogol cream — Apply at least two times a day on face, chest and upper arms during the 6 week treatment period
  Arms: cetomacrogol cream

SUMMARY:
Objective:

To assess the preemptive effect of Bepanthen® on decreasing the incidence of specific ≥ grade 2 dermatological side effects of interest in respect of compliance to EGFRI agents, HRQoL and the adherence during the 6-week skin treatment period. The adherence to the study creams will also be studied.

DETAILED DESCRIPTION:
Rationale:

Dermatological side effects, such as papulopustular eruption, xerosis, pruritus, periungual inflammation, mucosal-, and hair abnormalities, and edema occur in up to 90% of patients during treatment with epidermal growth factor receptor inhibitors (EGFRI). Patients are hindered in their daily activities and cannot maintain privacy about their illness because of the prominent side effects. The aesthetic discomfort, which is frequently associated with itching or painful skin or nails can lead to a decreased health related quality of life (HRQoL) and to dose reduction or discontinuation of anticancer treatment.

Patients with dermatological side effects have also an increased risk for cutaneous infections (at least 38%) which can complicate dermatological side effects.

At present, evidence of the effectiveness of the management options for dermatological side effects is lacking, and the effect of the dermatological side effects on HRQoL and adherence remains poorly understood.

Dexpanthenol cream (Bepanthen®, Bayer) has been used extensively to ameliorate acute radiation induced skin toxicity, diaper dermatitis, irritant hand dermatitis, graft-donor site wound healing and burn patients. The hypothesis is that its skin healing possibilities decreases this kind of side effects.

Study design:

Multicenter, two-arm randomized, double blind, prospective parallel group design, phase III study

Study population:

Each patient starting for the first time with EGFRI anticancer therapy which can cause papulopustular eruption (cetuximab, panitumumab, erlotinib, gefitinib, lapatinib, or other), will be included.

Intervention:

80 patients will receive for the first 6 weeks of treatment Bepanthen cream, 80 patients Cetomacrogol cream to apply twice daily. Using FACT-EGFRI, a dermatology-specific questionnaire, this study examines the effect of these side effects on three domains of HRQoL - symptoms, emotions, and functioning. Severity of dermatological side effects will be assessed using the NCI-CTCAE v4.0. Correlation of dermatology HRQoL scores with NCI-CTCAE grade, sex, age, type of EGFRI, and cancer type will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* ≥18 years of age.
* Patients must have signed an approved informed consent form prior to registration on study.
* Histological proof of cancer.
* A planned course of EGFRI treatment for any type of cancer. Patients must be entered on study ≤ 7 days before EGFRI treatment begins.
* Have an Eastern Co-operative Oncology Group (ECOG) performance status ≤ 2.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Patients need to be free of infection and not using any topical treatments on the skin.

Exclusion Criteria:

* Use of other concurrent topical creams or lotions at baseline.
* Concomitant use of medications that may affect trial results (e.a. concurrent use of topical antibiotics, topical steroids, and other topical treatments on face and chest within 14 days of Day 0 (baseline); treatment with any systemic antibiotics within 7 days prior to Day 0.
* Active dermatological conditions other than papulopustular eruption that may affect trial results. A skin examination reveals the presence of another skin disease in face or chest that may obscure rash to EGFRI and/or condition (excessive facial hair, excessive scarring, sunburn, or other disfigurement) located on the skin that, in the study physician's opinion, would confound the evaluation of the papulopustular eruption.
* Known allergy or hypersensitivity to ingredients in Bepanthen® or Cetomacrogol.
* Known sensitivity, papulopustular eruption or other abnormal skin reaction to topical or systemic medications or cleansing products at baseline.
* Prior treatment with targeted therapy of any kind.
* Current use of agents that are known to be strong inducers or inhibitors of CYP3A4 that can not be stopped

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-09; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
grade 2 or more papulopustular eruption | 6 weeks
  The incidence of grade ≥ 2 papulopustular eruption during the 6 week skin treatment within Bepanthen and Cetomacrogol, as measured by the CTCAE v4.0 and DERETT-H, an dermatologic specific healthcare provider questionnaire for Dermatological Reactions Targeted Therapy.
impact of papulopustular eruptions on HRQoL | 6 weeks
  Assess the impact of papulopustular eruptions on HRQoL as measured by the Functional Assessment of Cancer Therapy Questionnaire - EGFRI (FACT-EGFRI) and newly developed symptom experience diary Dermatological Reactions Targeted Therapy - Patients (DERETT-P).

SECONDARY OUTCOMES:
patient tolerability and satisfaction of study cream | 6 weeks
  Determine the patient tolerability and satisfaction of Bepanthen®/ Cetomacrogol cream as measured by DERETT-P.
effectiveness of study cream on the adherence | 6 weeks
  Determine the effectiveness of Bepanthen® cream versus Cetomacrogol cream on the adherence to anticancer agents as measured by FACT-EGFRI and DERETT-P.
other dermatological side effects | 6 weeks
  Assessments during the 6-week skin treatment period of the incidence and time to onset of other dermatological side effects which can appear together with papulopustular eruptions as measured by DERETT-H.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Boers-Doets, MSc, Study Chair — Waterland Hospital, Purmerend, the Netherlands; Mario Lacouture, MD, Principal Investigator — Memorial Sloan-Kettering Cancer Center, USA; Johan Nortier, PhD, Principal Investigator — Leiden University Medical Centre, the Netherlands
Locations (6):
- Netherlands (6):
  - Medisch Centrum Alkmaar, Alkmaar
  - Deventer ziekenhuis, Deventer
  - Admiraal de Ruyter Hospital, Goes
  - Leiden University Medical Centre, Leiden
  - Waterland Hospital, Purmerend
  - Zaans Medisch Centrum, Zaandam

REFERENCES:
- [Derived] Clabbers JMK, Boers-Doets CB, Gelderblom H, Stijnen T, Lacouture ME, van der Hoeven KJM, Kaptein AA. Xerosis and pruritus as major EGFRI-associated adverse events. Support Care Cancer. 2016 Feb;24(2):513-521. doi: 10.1007/s00520-015-2781-y. Epub 2015 Jun 27. PMID 26111953
- [Derived] Boers-Doets CB, Gelderblom H, Lacouture ME, Epstein JB, Nortier JW, Kaptein AA. Experiences with the FACT-EGFRI-18 instrument in EGFRI-associated mucocutaneous adverse events. Support Care Cancer. 2013 Jul;21(7):1919-26. doi: 10.1007/s00520-013-1752-4. Epub 2013 Feb 17. PMID 23417565